CLINICAL TRIAL: NCT01835444
Title: Worthy Assistants: Does Substituting Hospital Ward Care From Medical Residents to Physician Assistants Result in Cost Savings?
Brief Title: A Multicenter Research on the Effects of Substitution of Hospital Ward Care From Medical Doctors to Physician Assistants
Status: Completed | Type: Observational
Sponsor: Radboud University Medical Center (Other)
Collaborators: ZonMw: The Netherlands Organisation for Health Research and Development (Other)
Responsible Party: Sponsor
Other Study IDs: 80-82310-97-12094
Record Dates: First submitted 2013-04-05; First posted 2013-04-19 (Estimated); Last update posted 2015-05-14 (Estimated); Status verified 2015-05

CONDITIONS: Substitution of Care
Keywords: Physician Assistant; Substitution; Hospital ward care; Secondary health care

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- MD model: Hospital wards at which ward care is provided only by Medical Doctors (MDs)
- PA/MD model: Hospital wards at which ward care is provided by both Physician Assistants (PAs) and Medical Doctors (MDs)
  Interventions: Other: PA/MD model

INTERVENTIONS:
Other: PA/MD model — Intervention wards are hospital wards at which ward care is provided by both Physician Assistants (PAs) and Medical Doctors (MDs)
  Groups: PA/MD model

SUMMARY:
Reallocation of healthcare is one solution to the problems healthcare is facing. In the Netherlands reallocation of care to Physician Assistants (PAs) hasn't adequately been studied. Given the growing number of PAs, it is essential to evaluate the effectiveness and efficacy of (Dutch) PA services.

This multicenter matched-controlled study aims to evaluate the (cost) effectiveness of substitution of hospital ward care from medical doctors (MDs) to PAs. The traditional model in which the role of house officer is taken by medical doctors MD model) will be compared with a mixed model in which a PA functions as house officer together with a medical doctor (PA/MD model). Hospital wards will be matched on medical specialism and hospital type (i.e. academic;non-academic). On the basis of USA studies, it is hypothesized that the mixed PA/MD model compared to the MD model reduces the costs of healthcare, while improving or maintaining the clinical outcomes, patients and provider satisfaction, and continuity and quality of care.

Primary research question:

• What is the effect of 'mixed PA/MD model' compared with 'MD model' on efficiency of care?

Secondary research questions:

* What is the effect of 'mixed PA/MD model' compared with 'MD model' on clinical and patients outcomes?
* What is the effect of 'mixed PA/MD model' compared with 'MD model' on continuity of care?
* What is the effect of 'mixed PA/MD model' compared with 'MD model' on nurses and (specialist) medicals doctor experiences?
* What are the barriers and facilitating factors considering the implementation of PAs as house officer?

ELIGIBILITY:
Inclusion criteria:

• Wards using a mixed PA/physician model (with PA ward coverage of at least 50% of the available ward hours per week, during dayshifts on weekdays) or a physician model (daily coverage by a (specialized medical doctor)

Exclusion criteria on ward level:

* Wards from specialty hospitals
* Wards with only PAs in training
* Wards with a nurse practitioner (NP) in the role of house officer (NP, NP/MD or PA/NP/MD model)
* Pediatric and psychiatric wards, intensive care units

Exclusion criteria on patient level:

* Terminal patients
* Not fluent in Dutch language
* Age < 18 years
* Patients in daycare

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Hospital Ward Care: all patients (age 18 years or older) admitted to a hospital ward will be included in the study.
Sampling Method: Non-Probability Sample
Enrollment: 2382 (Actual)
Dates: Start 2013-04; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Length of hospital stay | Patients will be followed for the duration of hospital stay; an expected average of 6 days
  The difference between date of discharge and date of admission

SECONDARY OUTCOMES:
Efficiency of care | Patients will be followed from hospital admission till 1 month after discharge; an expected average of 1 month and 6 days
  Relevant costs associated with the principal admission (length of hospital stay, resource use, consultation of health care suppliers, salaries) and costs that occurred after discharge (unplanned readmission, presentation at emergency departments, visits of general practitioner, required home care) will be calculated, considering a follow-up period from admission until 1 month after discharge. All volumes will be collected in detail at an individual patient level, primarily from medical patient records and patient and care provider questionnaires. Medical costs will be calculated by multiplying the volumes of healthcare use with corresponding unit prices, derived from the Dutch Manual for Costing Research
Quality of hospital ward care | Patients will be followed from hospital admission till 1 month after discharge; an expected average of 1 month and 6 days
  To estimate the quality of ward care, a set of objective indicators has been developed through literature review and clinical input from a physician panel. We have selected both clinical indicators and process indicators, with a follow-up period of maximum 1 month after discharge. Clinical indicators were based on the national set of indicators for quality of hospital care from the Dutch Health Care Inspectorate (IGZ) and consider the incidences of inhospital mortality, cardiopulmonary resuscitation, unplanned readmission, presentation at emergency department after discharge,unplanned transfer to Intensive Care Unit, development of hospital infections, pressure sore and fever, and pain scores . Process indicators are the number of days between a patients discharge and the date of written turnover to general practitioner or other hospital, and acquaintance with the patient within 24 hours after admission
Patient quality of life | Patients will be followed from hospital admission till 1 month after discharge; an expected average of 1 month and 6 days. Measurements of quality of life will be performed at hospital admission, hospital discharge and 1 month after discharge
  Patient experienced quality of life will be measured by the EQ-5D questionnaire. This questionnaire will be distributed at hospital admission, hospital discharge, and 1 month after discharge
Feasibility, barriers and facilitators | 12 months
  Semi-structured (group)interviews will be held with PAs, (specialized) medical doctors, ward nurses and heads of the departments. The interviews will cover experiences with the utilized ward model, communication between professionals, satisfaction, and barriers and facilitators related to the utilization of the 'mixed PA/MD model'. Specific attention will be paid to the role and functioning of PAs
Care provider experiences | 12 months
  Job satisfaction, subjective workload and stress reaction of PAs, (specialized) medical doctors and ward nurses will be measured by a self-administered questionnaire. Job satisfaction will be measured by an adapted version of the job satisfaction questionnaire of McCranie, stress reaction will be measured by a short version of the General Health Questionnaire (GHQ-12)
  Objective workload will be measured by calculating the ratio between number of working hours at the hospital ward, and the number of patients the PA or medical doctor is responsible for.
Continuity of care | 4 months
  Continuity of care will be measured by deriving the number of rotations of PAs and medical doctors at the hospital ward from work schedules, which will be assessed during 4 weeks, spread over 4 months
Patient experiences with hospital ward care | Patients will be followed for the duration of hospital stay; an expected average of 6 days. Measurement of patient experiences will be performed at discharge
  Patient experiences with medical ward care will be assessed by a self-administered questionnaire at discharge. This questionnaire focuses on satisfaction with communication, experienced continuity of care and cooperation, and the patients view on the medical competencies of the ward care provider

CONTACTS AND LOCATIONS:
Overall Officials: M.G.H. Laurant, PhD, Principal Investigator — IQ healthcare, UMC St Radboud
Locations (23):
- Netherlands (23):
  - Scheper Ziekenhuis, Emmen, Drenthe
  - Gelre Ziekenhuizen, Apeldoorn, Gelderland
  - Rijnstate, Arnhem, Gelderland
  - Slingeland Ziekenhuis, Doetinchem, Gelderland
  - Ziekenhuis de Gelderse Vallei, Ede, Gelderland
  - Radboud University Nijmegen Medical Centre, Nijmegen, Gelderland
  - Canisius Wilhelmina ziekenhuis, Nijmegen, Gelderland
  - Streekziekenhuis Koningin Beatrix, Winterswijk, Gelderland
  - Laurentius Ziekenhuis, Roermond, Limburg
  - Orbis Medisch Centrum, Sittard, Limburg
  - VieCuri Medical Center, Venlo, Limburg
  - Jeroen Bosch Ziekenhuis, 's-Hertogenbosch, North Brabant
  - Lievensberg Ziekenhuis, Bergen op Zoom, North Brabant
  - Elkerliek ziekenhuis, Helmond, North Brabant
  - Fransiscus Ziekenhuis, Roosendaal, North Brabant
  - St. Elisabeth Ziekenhuis, Tilburg, North Brabant
  - TweeSteden Ziekenhuis, Tilburg, North Brabant
  - Tjongerschans ziekenhuis, Heerenveen, Provincie Friesland
  - Reinier de Graaf Gasthuis, Delft, South Holland
  - HagaZiekenhuis, The Hague, South Holland
  - Medisch Centrum Haaglanden, The Hague, South Holland
  - UMC Utrecht, Utrecht, Utrecht
  - Van Weel Bethesda Ziekenhuis, Dirksland, Zeeland

REFERENCES:
- [Derived] Timmermans MJC, van Vught AJAH, Peters YAS, Meermans G, Peute JGM, Postma CT, Smit PC, Verdaasdonk E, de Vries Reilingh TS, Wensing M, Laurant MGH. The impact of the implementation of physician assistants in inpatient care: A multicenter matched-controlled study. PLoS One. 2017 Aug 9;12(8):e0178212. doi: 10.1371/journal.pone.0178212. eCollection 2017. PMID 28793317
- [Derived] Timmermans MJC, van den Brink GT, van Vught AJAH, Adang E, van Berlo CLH, Boxtel KV, Braunius WW, Janssen L, Venema A, van den Wildenberg FJ, Wensing M, Laurant MGH. The involvement of physician assistants in inpatient care in hospitals in the Netherlands: a cost-effectiveness analysis. BMJ Open. 2017 Jul 10;7(7):e016405. doi: 10.1136/bmjopen-2017-016405. PMID 28698344
- [Derived] Timmermans MJ, van Vught AJ, Van den Berg M, Ponfoort ED, Riemens F, van Unen J, Wobbes T, Wensing M, Laurant MG. Physician assistants in medical ward care: a descriptive study of the situation in the Netherlands. J Eval Clin Pract. 2016 Jun;22(3):395-402. doi: 10.1111/jep.12499. Epub 2015 Dec 23. PMID 26695837
- [Derived] Timmermans MJ, van Vught AJ, Wensing M, Laurant MG. The effectiveness of substitution of hospital ward care from medical doctors to physician assistants: a study protocol. BMC Health Serv Res. 2014 Jan 28;14:43. doi: 10.1186/1472-6963-14-43. PMID 24472112